CLINICAL TRIAL: NCT02708784
Title: Function, Structure and Quality of Striated Muscles in Patients With Muscular Diseases - an MRI Study on Pompe Disease and Dystrophia Myotonica
Brief Title: An MRI Study on Muscular Diseases -Pompe Disease and Dystrophia Myotonica-
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: PsDM15RMBH
Record Dates: First submitted 2015-12-08; First posted 2016-03-15 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2015-11

CONDITIONS: Glycogen Storage Disease Type 2; Dystrophia Myotonica
Keywords: Glykogen storage disease type 2); Dystrophia Myotonica; Muscular disorders; MR-imaging; Muscle strength; Myopathies
MeSH Terms: conditions — Glycogen Storage Disease Type II; Myotonic Dystrophy; Muscular Diseases

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Pompe disease: Patients will perform muscle strength measurement with dynamometer and MR-imaging. After 8 months the investigations will be repeated.
- Myotonic Dystrophy: Patients will perform muscle strength measurement with dynamometer and MR-imaging. The investigations will not be repeated after 8 months.
- Healthy controls: Patients will perform muscle strength measurement with dynamometer and MR-imaging. The investigations will not be repeated after 8 months.

SUMMARY:
The aim of the project is to develop new Magnetic Resonance (MR) imaging techniques for better diagnosis and monitoring of patients with muscular disorders.

Muscle quality in patients with Late Onset Pompe Disease (Acid Maltase Deficiency type 2) and in patients with Myotonica Dystrophy will be evaluated, by determining muscle strength in relation to muscle size and muscle strength in relations to fat-muscle ratio.

DETAILED DESCRIPTION:
The investigators focus on the rare Glycogen Storage Disease type 2 (Pompe Disease), a genetic disease characterized by gradual replacement of muscular tissue with glycogen and fat, resulting in loss of muscle mass and muscle strength. Pompe disease is of particular interest since a new drug has recently been developed and approved for this, hitherto untreatable, condition. This treatment is expensive, and it is therefore of great importance to have objective methods of examination to monitor the disease and the effects of the treatment.

Until now, monitoring has been based primarily on physical test such as the 6 min walking test and isokinetic dynamometry. These methods may not be sensitive enough to detect changes for shorter periods in slowly progressing-diseases. New MRI techniques may be useful for monitoring in myopathies.

The other disease the investigators are focusing on is Myotonic Dystrophy, because of its great similarities with Pompe Disease. As with Pompe disease, the muscular tissue slowly degenerate and fat infiltrations occur.

Hypothesis

In this study, the investigators want to test the following hypotheses:

* Intrinsic muscle strength in patients with Pompe disease and Myotonic Dystrophy is linear correlated with muscle to fat volume ratios from MR images.
* Disease grade in patients with Pompe disease and Myotonic Dystrophy corresponds to the extent of fat proliferation in the muscles of the lower extremities.
* Intrinsic muscle strength is a more specific and sensitive method to reveal the effects of enzyme replacement treatment in patients with Pompe than the 6 minutes-walking-test.

Methods Fifteen patients with LOPD from Denmark and from Germany (Münster), 15 patients with Myotonic Dystrophy and 30 controls are included.

The MR protocol includes the special T1 weighted sequence DIXON (1x1x3mm3; TR: 5.31ms TE: 2.46ms) enabling acquisition of muscle and fat images at 3 Tesla (Magnetom-Skyra, Siemens AG, Erlangen, Germany). The MR scans will consist of 400 axial slices covering from L1 to the ankle resulting in a total scan time of 22½ minutes.

Muscle strength will be measured by isokinetic dynamometry. The measurement will be done using the Biodex System 3 PRO Dynamometer (Biodex Medical Systems Inc. NY, USA) for which a standardized protocol has been developed.

Maximal isokinetic strength of extensors and flexors of the dominating arm and extensor and flexors at the knee, ankle and hip of the non-dominant lower extremity will be measured.

There are no known side effects related to MR-scanning. During the examination, the subjects will wear headphones in order to reduce the high sounds that come from the scanning machine. The scan is painless and there is no use of contrast. The only disadvantage is that the person has to lie motionless for 20-30 minutes. There are some security rules to respect in order to avoid accidents due to metals being attracted by the machine's strong magnetic field.

No side effects are associated to muscle strength measurement with the Dynamometer.

However, weak patients may be a bit tired after the examination, as they have to perform some movements using all their force.

Statistics Comparison between baseline and visits will be performed using conventional statistic methods as unpaired t-test or non-parametric tests such as Wilcoxon signed-rank test. In variation analyses of several groups ANOVA and ANCOVA will be used. A significant difference of p-values below 0.05 has to be determined, to determine the validity of the findings. With a significant level of 5% a power calculation estimated a needed sample size of 14 patients, with a power of 90%. The calculation is based on an expected decrease in muscle volume compared to fat (1.2 vs 0.95 with a standard deviation of 0.2). The power calculation is an estimate, but compared to a similar studyxiii the sample size includes an extra 3 subjects. Given the rare condition of PD, inclusion of patients will continue even if the required minimum is not achieved.

The same statistics calculation will be used for patients with Dystrophia Myotonica, who are included in the study because of its great similarities with Pompe Disease.

Perspectives If MRI imaging is a sensitive method with high specificity for the assessment of muscle quality in myopathies, this technique may be used for diagnosis and continuous validation of the proper treatment of patients with Pompe disease and with related muscular diseases.

Clinical trial: Day one. Patients with Pompe Disease and Dystrophia Myotonica The patients will come to the neurological department of Aarhus University Hospital at Nørrebrogade. Their muscle-strength will be measured by the Dynamometer; these measurements will take approximately 2 hours.

In addition, Pompe patients will undergo the 6 min walking test, the vital capacity and negative inspiration/expiration tests, the sit-to-stand test as well as a structured neurological examination. This will take about 1 hour.

After the first part of the examinations, the patients will be driven, by the hospital minibus, to the MR center at Skejby University Hospital, where the MR-scanning will be done. The total timeframe for the scanning, included change of clothes, information and scanning, will take 1,5 hours. In case that it´s not possible to make the physical examinations and the scanning on the same day, the scanning will take place another day, within the following 7 working days.

Healthy controls The control subjects will be received at the neurological department of Aarhus University Hospital at Nørrebrogade. Their muscle-strength will be measured by the Dynamometer; the measurements will take approximately 2 hours. Afterwards, they will be driven, by the hospital minibus, to the MR center at Skejby University Hospital, where the MR-scanning will be performed. The total time for the scanning, included changes of clothes, information and scanning, will take 1,5 hours. In case that it´s not possible to perform both the physical examinations and the scanning on the same day, the scanning will take place another day, within the following 7 working days.

Clinical trial: day 2 After 8 months, patients with Pompe disease will come for new investigations. The same examinations, as described above, will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed Pompe disease patients, whether they are in treatment with ERT or not, or Diagnosed Dystrophia Myotonica patients.
* Healthy controls, have to be sex and age-matched to patients with muscular disease.

Exclusion Criteria:

* Age under 18 years.
* The subjects must be able to perform an MR-scanning. Moreover they have to sign and respect the MR security rules "Kontrol skema før MR undersøgelse" and "Patient information i forbindelse med MR scanning".
* The subjects must be capable of performing the muscle strength test by the Dynamometer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited trough their attendance to the Hospital. Pompe disease patients will be recruited from all the treating hospitals in Denmark and from the University hospital of Münster. Patients with Myotonic Dystrophy will be recruited trough their attendance at Aarhus University Hospital.
  Healthy controls will be recruited from the general Danish population.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-08 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Muscle strength in Newton*meter | one year
  Muscle strength in measured by dynamometry, and the used outcome is the "peak torque".
Muscle to fat ratio | one year
  Calculated from the MR-images, is a measure for muscle quality. The calculations are based on the signal intensity of the fat and water Dixon MR-images.
Volume ratio | one year
  Defined from the MR-images, is a measure for muscle quality.

SECONDARY OUTCOMES:
6 minutes walking test | one year
  Only for Pompe disease participants
Forced Vital Function | on year
  Only for Pompe disease participants

CONTACTS AND LOCATIONS:
Overall Officials: Henning Andersen, Professor, Study Chair — Aarhus University Hospital
Locations (2):
- Denmark (2):
  - Department of Neurology, Aarhus University Hospital, Aarhus C
  - MR centre, Skejby University Hospital., Aarhus N

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ausems MG, Verbiest J, Hermans MP, Kroos MA, Beemer FA, Wokke JH, Sandkuijl LA, Reuser AJ, van der Ploeg AT. Frequency of glycogen storage disease type II in The Netherlands: implications for diagnosis and genetic counselling. Eur J Hum Genet. 1999 Sep;7(6):713-6. doi: 10.1038/sj.ejhg.5200367. PMID 10482961
- [Background] van der Ploeg AT, Reuser AJ. Pompe's disease. Lancet. 2008 Oct 11;372(9646):1342-53. doi: 10.1016/S0140-6736(08)61555-X. PMID 18929906
- [Background] Hagemans ML, Winkel LP, Van Doorn PA, Hop WJ, Loonen MC, Reuser AJ, Van der Ploeg AT. Clinical manifestation and natural course of late-onset Pompe's disease in 54 Dutch patients. Brain. 2005 Mar;128(Pt 3):671-7. doi: 10.1093/brain/awh384. Epub 2005 Jan 19. PMID 15659425
- [Background] van der Ploeg AT, Clemens PR, Corzo D, Escolar DM, Florence J, Groeneveld GJ, Herson S, Kishnani PS, Laforet P, Lake SL, Lange DJ, Leshner RT, Mayhew JE, Morgan C, Nozaki K, Park DJ, Pestronk A, Rosenbloom B, Skrinar A, van Capelle CI, van der Beek NA, Wasserstein M, Zivkovic SA. A randomized study of alglucosidase alfa in late-onset Pompe's disease. N Engl J Med. 2010 Apr 15;362(15):1396-406. doi: 10.1056/NEJMoa0909859. PMID 20393176
- [Background] Toscano A, Schoser B. Enzyme replacement therapy in late-onset Pompe disease: a systematic literature review. J Neurol. 2013 Apr;260(4):951-9. doi: 10.1007/s00415-012-6636-x. Epub 2012 Aug 28. PMID 22926164
- [Background] Anderson LJ, Henley W, Wyatt KM, Nikolaou V, Waldek S, Hughes DA, Lachmann RH, Logan S. Effectiveness of enzyme replacement therapy in adults with late-onset Pompe disease: results from the NCS-LSD cohort study. J Inherit Metab Dis. 2014 Nov;37(6):945-52. doi: 10.1007/s10545-014-9728-1. Epub 2014 Jun 7. PMID 24906254
- [Background] Mercuri E, Pichiecchio A, Allsop J, Messina S, Pane M, Muntoni F. Muscle MRI in inherited neuromuscular disorders: past, present, and future. J Magn Reson Imaging. 2007 Feb;25(2):433-40. doi: 10.1002/jmri.20804. PMID 17260395
- [Background] Ponrartana S, Ramos-Platt L, Wren TA, Hu HH, Perkins TG, Chia JM, Gilsanz V. Effectiveness of diffusion tensor imaging in assessing disease severity in Duchenne muscular dystrophy: preliminary study. Pediatr Radiol. 2015 Apr;45(4):582-9. doi: 10.1007/s00247-014-3187-6. Epub 2014 Sep 23. PMID 25246097
- [Background] Carlier RY, Laforet P, Wary C, Mompoint D, Laloui K, Pellegrini N, Annane D, Carlier PG, Orlikowski D. Whole-body muscle MRI in 20 patients suffering from late onset Pompe disease: Involvement patterns. Neuromuscul Disord. 2011 Nov;21(11):791-9. doi: 10.1016/j.nmd.2011.06.748. Epub 2011 Jul 30. PMID 21803581
- [Background] Pichiecchio A, Uggetti C, Ravaglia S, Egitto MG, Rossi M, Sandrini G, Danesino C. Muscle MRI in adult-onset acid maltase deficiency. Neuromuscul Disord. 2004 Jan;14(1):51-5. doi: 10.1016/j.nmd.2003.08.003. PMID 14659413
- [Background] Vielhaber S, Brejova A, Debska-Vielhaber G, Kaufmann J, Feistner H, Schoenfeld MA, Awiszus F. 24-months results in two adults with Pompe disease on enzyme replacement therapy. Clin Neurol Neurosurg. 2011 Jun;113(5):350-7. doi: 10.1016/j.clineuro.2010.09.016. Epub 2011 Apr 7. PMID 21477922
- [Background] Alejaldre A, Diaz-Manera J, Ravaglia S, Tibaldi EC, D'Amore F, Moris G, Muelas N, Vilchez JJ, Garcia-Medina A, Uson M, Martinez Garcia FA, Illa I, Pichiecchio A. Trunk muscle involvement in late-onset Pompe disease: study of thirty patients. Neuromuscul Disord. 2012 Oct 1;22 Suppl 2:S148-54. doi: 10.1016/j.nmd.2012.05.011. PMID 22980766
- [Background] Pichiecchio A, Poloni GU, Ravaglia S, Ponzio M, Germani G, Maranzana D, Costa A, Repetto A, Tavazzi E, Danesino C, Moglia A, Bastianello S. Enzyme replacement therapy in adult-onset glycogenosis II: is quantitative muscle MRI helpful? Muscle Nerve. 2009 Jul;40(1):122-5. doi: 10.1002/mus.21304. PMID 19533640
- [Background] Ravaglia S, Pichiecchio A, Ponzio M, Danesino C, Saeidi Garaghani K, Poloni GU, Toscano A, Moglia A, Carlucci A, Bini P, Ceroni M, Bastianello S. Changes in skeletal muscle qualities during enzyme replacement therapy in late-onset type II glycogenosis: temporal and spatial pattern of mass vs. strength response. J Inherit Metab Dis. 2010 Dec;33(6):737-45. doi: 10.1007/s10545-010-9204-5. Epub 2010 Sep 16. PMID 20844963
- [Background] Andreassen CS, Schlutter JM, Vissing J, Andersen H. Effect of enzyme replacement therapy on isokinetic strength for all major muscle groups in four patients with Pompe disease-a long-term follow-up. Mol Genet Metab. 2014 May;112(1):40-3. doi: 10.1016/j.ymgme.2014.02.015. Epub 2014 Mar 5. PMID 24685124
- [Background] Hiba B, Richard N, Hebert LJ, Cote C, Nejjari M, Vial C, Bouhour F, Puymirat J, Janier M. Quantitative assessment of skeletal muscle degeneration in patients with myotonic dystrophy type 1 using MRI. J Magn Reson Imaging. 2012 Mar;35(3):678-85. doi: 10.1002/jmri.22849. Epub 2011 Nov 8. PMID 22069222